CLINICAL TRIAL: NCT00219609
Title: A Phase 2 Multi-Center, Open Label Long-Term Extension Trial To Assess The Safety Of Oral Uk-390,957 Administered As Required In Adult Men With Premature Ejaculation
Brief Title: Assessment Of Safety Of UK-390,957
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3871028
Record Dates: First submitted 2005-09-09; First posted 2005-09-22 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Ejaculation

INTERVENTIONS:
Drug: UK-390,957

SUMMARY:
To determine whether UK-390,957 is a safe treatment for premature ejaculation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have completed one of the phase 2 trials (A3871022/ A3871027/ A3871029) and will have met the diagnostic criteria for premature ejaculation as defined by DSM-IV

Exclusion Criteria:

* No drug related serious adverse events

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1058
Dates: Start 2005-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Assessment of safety

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (82):
- United States (46):
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Atherton, California
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Laguna Woods, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Redwood City, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Tarzana, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Saint Clair Shores, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Southhaven, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Edison, New Jersey
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Vorhees, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, West Seneca, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, Milwuakee, Wisconsin
- Australia (5):
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Spring Hill, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Malvern, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia
- Austria (2):
  - Pfizer Investigational Site, Mistelbach
  - Pfizer Investigational Site, Salzburg
- Canada (6):
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, MontrÃ©al, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
- Czechia (2):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Prague
- Pfizer Investigational Site, Lyon, France
- Germany (3):
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, München
- Israel (4):
  - Pfizer Investigational Site, Beersheba
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, Tel Aviv
  - Pfizer Investigational Site, Tel Litwinsky
- Italy (2):
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Roma
- Norway (2):
  - Pfizer Investigational Site, Moelv
  - Pfizer Investigational Site, Oslo
- Poland (2):
  - Pfizer Investigational Site, Mysłowice
  - Pfizer Investigational Site, Warsaw
- Sweden (2):
  - Pfizer Investigational Site, Skövde
  - Pfizer Investigational Site, Stockholm
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Balcali, Adana
  - Pfizer Investigational Site, Samanpazarı, Ankara
  - Pfizer Investigational Site, Balçova, İzmir
- United Kingdom (2):
  - Pfizer Investigational Site, Nr Lichfield, Staffordshire
  - Pfizer Investigational Site, Devon

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3871028&StudyName=Assessment+Of+Safety+Of+UK%2D390%2C957